CLINICAL TRIAL: NCT03584152
Title: Postoperative Pain Management in Rhinoplasty: A Randomized Controlled Trial
Brief Title: Postoperative Pain Management in Rhinoplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sam P. Most, Chief, Division of Facial Plastic and Reconstructive Surgery, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 46945
Record Dates: First submitted 2018-06-27; First posted 2018-07-12 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Pain, Postoperative
Keywords: Postoperative pain; Rhinoplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — oxycodone-acetaminophen; acetaminophen, hydrocodone drug combination; Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Drug Arm A (Active Comparator): Norco 5mg-325 mg Tablet, administered orally every 4 hours for 5 days total
  Interventions: Drug: Norco 5Mg-325Mg Tablet
- Drug Arm B (Active Comparator): Tylenol 325 mg Caplet, administered orally every 4 hours for 5 days total. Ibuprofen 200 mg administered orally every 4 hours for 5 days total.
  Interventions: Drug: Tylenol 325Mg Caplet; Drug: Ibuprofen 200 mg

INTERVENTIONS:
Drug: Norco 5Mg-325Mg Tablet — Opioid Analgesics
  Other Names: Lortab; Vicodin; Hycet
  Arms: Drug Arm A
Drug: Tylenol 325Mg Caplet — Non opioid analgesics
  Other Names: Acetaminophen
  Arms: Drug Arm B
Drug: Ibuprofen 200 mg — Non opioid analgesics
  Other Names: Advil; Motrin
  Arms: Drug Arm B

SUMMARY:
The primary purpose of the study is to determine adequacy of postoperative pain control after nasal surgery in patients prescribed Acetaminophen (325mg) + Hydrocodone (5mg) compared to Acetaminophen(325mg) + Ibuprofen (200mg)for a period of 5 days after nasal surgery. To assess the degree of pain, the participants will score the intensity of their pain on a visual analog scale(VAS)of 0-100points (0- no pain and 100- most severe pain), preoperatively and postoperatively (to be documented before each dose) for the duration of the prescribed medications .

Additionally, the study will also seek to track:

1. The total number of pills each patients consume from the prescribed 5 day regimen.
2. Any associated side effects.
3. Additional pain medications prescribed in case of inadequate pain control, postoperatively.

DETAILED DESCRIPTION:
From this study, the investigators hope to learn the following:

1. Is adequate postoperative pain management after nasal surgery achieved with opioid or non-opioid drugs?
2. If opioid drugs are required for adequate pain control postoperatively, is it possible to reduce the number of days the drugs are prescribed for?
3. What are the common side effect profiles of the included drugs?

In light of the current opioid epidemic in the country, it is important the the physicians explore the utility of drugs other than opioids for adequate postoperative pain management. Also, reducing the dosage and/or number of prescribed opioid drugs lessens the propensity for misuse of physician prescribed opioid medications.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Able to speak and understand english.
* Undergoing rhinoplasty for cosmetic purposes
* Undergoing rhinoplasty for treatment of nasal obstruction

Exclusion Criteria:

* Less than 18 years of age
* Cannot speak and understand english
* Patients who have undergone nasal surgery in the past
* Patients not undergoing nasal surgery
* Women will be excluded if they are either pregnant or lactating as this population does not undergo nasal surgery at our center.
* Patients with any known allergies to the class of pain medications used in the study.

Please note: Any person interested in this clinical trial should contact the Facial Plastic and Reconstructive Surgery clinic at (650) 736 - 3223 to schedule a consultation with Dr. Sam P. Most to assess their eligibility for the trial. Please note, enrolling in the clinical trial will not entitle the participant to a waiver of charges associated with undergoing nasal surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2025-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SAM P Most, MD, Principal Investigator — Stanford University
Locations (1):
- Facial Plastic and Reconstructive Surgery Clinic, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Johns MD. Transfer of a pattern versus component discrimination following training in a probabilistic situation. J Exp Psychol. 1965 Nov;70(5):506-9. doi: 10.1037/h0022535. No abstract available. PMID 5833672

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from the day of the pre-operative appointment (approximately 2 to 4 weeks prior to procedure) through post-operative day 7. Follow-up data at two time points (<6 months, and ≥ 6 months) were obtained by chart review.
Pre-assignment Details: 159 signed informed consent and 141 participants were randomized.
Period: Overall Study
Arm/Group | Drug Arm A | Drug Arm B
Started | 72 | 69
Completed | 65 | 65
Not Completed | 7 | 4
Not completed — Discontinued intervention | 7 | 4

BASELINE CHARACTERISTICS:
Population: Participants who completed the intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug Arm A | Drug Arm B | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (8.6) | 33.5 (12.4) | 32.1 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 52 | 100
  Male | 17 | 13 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 44 | 45 | 89
  Asian | 15 | 10 | 25
  Latino/ Hispanic | 6 | 10 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 65 | 65 | 130

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Visual Analog Scale (VAS)- 0-100 (0- no Pain and 100- Most Severe Pain)
Description: Self reported pain intensity at every prescribed dose averaged over a period of 5 days.
Time Frame: 5 days post-operative [up to approximately 5 weeks post-baseline]
Population: Participants who completed the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Drug Arm A | Drug Arm B
Number analyzed (Participants) | 65 | 65
score on a scale | 44 (14.1) | 41 (16.3)
Statistical Analysis 1: Comparison: Drug Arm A vs Drug Arm B; Test type: Non-Inferiority — The null hypothesis stated that the combination of treatment arm B is worse than the combination of treatment arm A by more than -Δ, where -Δ is the 'non-inferiority margin.'; p = 0.156, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05

2. Secondary Outcome: Number of Study Drugs (Doses) Utilized
Description: Use of any study medication, excluding tramadol.
Time Frame: 5 days
Population: Participants who completed the intervention.
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Drug Arm A | Drug Arm B
Number analyzed (Participants) | 65 | 65
doses | 16 (9.5) | 19 (9.9)
Statistical Analysis 1: Comparison: Drug Arm A vs Drug Arm B; Test type: Other; p = 0.112, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05

3. Secondary Outcome: Number of Tramadol Doses Utilized
Time Frame: 5 days
Population: Participants who completed the intervention.
Measure: Mean (Standard Deviation); unit: doses
Arm/Group | Drug Arm A | Drug Arm B
Number analyzed (Participants) | 65 | 65
doses | 1 (2.5) | 2.0 (3.7)
Statistical Analysis 1: Comparison: Drug Arm A vs Drug Arm B; Test type: Other; p = 0.803, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05

4. Secondary Outcome: Number Patients Who Reported Adequate Pain Control
Time Frame: 5 days
Population: Participants who completed the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Arm A | Drug Arm B
Number analyzed (Participants) | 65 | 65
Participants
  No (not adequate) | 4 | 2
  Yes (adequate) | 61 | 63
Statistical Analysis 1: Comparison: Drug Arm A vs Drug Arm B; Test type: Other; p = 0.403, Chi-squared — The a priori threshold for statistical significance was < 0.05

5. Secondary Outcome: Side Effects of Pain Medications
Description: Self reported side effects of prescribed medications according to response options. Participants may have reported more than one side-effect. Commonly experienced medication side-effects would not necessarily be considered to be adverse events.
Time Frame: 5 days
Population: Participants who completed the intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Drug Arm A | Drug Arm B
Number analyzed (Participants) | 65 | 65
Participants
  Nausea | 17 | 13
  Itchiness | 14 | 2
  Constipation | 22 | 19
  Dizziness | 41 | 31
  Bleeding | 30 | 28
  Headache | 9 | 8
  Other | 7 | 3
Statistical Analysis 1: Comparison: Drug Arm A vs Drug Arm B; Difference between-groups in nausea; Test type: Other; p = 0.405, Chi-squared — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: Drug Arm A vs Drug Arm B; Difference between-groups in itchiness; Test type: Other; p = 0.001, Fisher Exact — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 3: Comparison: Drug Arm A vs Drug Arm B; Difference between-groups in constipation; Test type: Other; p = 0.571, Chi-squared — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 4: Comparison: Drug Arm A vs Drug Arm B; Difference between-groups in dizziness; Test type: Other; p = 0.078, Chi-squared — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 5: Comparison: Drug Arm A vs Drug Arm B; Difference between-groups in bleeding; Test type: Other; p = 0.724, Chi-squared — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 6: Comparison: Drug Arm A vs Drug Arm B; Difference between-groups in headache; Test type: Other; p = 0.795, Chi-squared — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 7: Comparison: Drug Arm A vs Drug Arm B; Difference between-groups in "other" side effects; Test type: Other; p = 0.188, Fisher Exact — The a priori threshold for statistical significance was < 0.05

6. Secondary Outcome: Standardized Cosmesis and Health Nasal Outcomes Survey (SCHNOS) Questionnaire
Description: The SCHNOS-O (obstructive) and SCHNOS-C (Cosmesis) scores were rated from 0 to 100 (higher scores correspond to worse obstruction or cosmesis). Not all 130 patients had a postoperative score at both time follow-up intervals (<6 months, and ≥ 6 months, obtained by chart review), thus a mean postoperative score (SD) was calculated for each treatment group accounting for both intervals.
Time Frame: Baseline and post-operative follow-up (up to an average of 12 months following procedure)
Population: Participants who completed the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Drug Arm A | Drug Arm B
Number analyzed (Participants) | 65 | 65
score on a scale
  SCHNOS-O (pre-operative) | 40.0 (33.2) | 41.0 (36.1)
  Change in SCHNOS-O (post-operative) | -25.7 (35.0) | -23.4 (41.9)
  SCHNOS-C (pre-operative) | 54.0 (29.0) | 54.0 (26.4)
  Change in SCHNOS-C (post-operative) | -39.6 (30.7) | -36.0 (34.2)
Statistical Analysis 1: Comparison: Drug Arm A vs Drug Arm B; Difference in change in SCHNOS-O; Test type: Other; p = 0.7318, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: Drug Arm A vs Drug Arm B; Difference in change in SCHNOS-C; Test type: Other; p = 0.5267, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05

7. Secondary Outcome: Visual Analog Scale-Functional (VAS-F)
Description: Patient's perceived severity of their nasal obstruction was self-graded using a 10-cm-long visual analogue scale ('0' indicated 'no nasal obstruction' and '10' indicated 'worst possible nasal obstruction). Not all 130 patients had a postoperative score at both time follow-up intervals (<6 months, and ≥ 6 months, obtained by chart review), thus a mean postoperative score (SD) was calculated for each treatment group accounting for both intervals.
Time Frame: Baseline and post-operative follow-up (up to an average of 12 months following procedure)
Population: Participants who completed the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Drug Arm A | Drug Arm B
Number analyzed (Participants) | 65 | 65
score on a scale
  Pre-operative | 4.0 (3.1) | 4.0 (3.1)
  Post-operative (change) | -1.8 (3.0) | -1.8 (3.5)
Statistical Analysis 1: Comparison: Drug Arm A vs Drug Arm B; Difference in change in VAS-F; Test type: Other; p = 0.9158, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05

8. Secondary Outcome: Visual Analog Scale-Aesthetic (VAS-A)
Description: Patient's perceived aesthetic appearance was self-graded using a 10-cm-long visual analogue scale ('0' indicated 'completely dissatisfied with nasal appearance' and '10' indicated 'the highest possible satisfaction with nasal appearance'). Not all 130 patients had a postoperative score at both time follow-up intervals (<6 months, and ≥ 6 months, obtained by chart review), thus a mean postoperative score (SD) was calculated for each treatment group accounting for both intervals.
Time Frame: Baseline and post-operative follow-up (up to an average of 12 months following procedure)
Population: Participants who completed the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Drug Arm A | Drug Arm B
Number analyzed (Participants) | 65 | 65
score on a scale
  Pre-operative | 3.0 (2.3) | 3.0 (2.5)
  Post-operative (change) | -1.5 (2.7) | -1.2 (3.1)
Statistical Analysis 1: Comparison: Drug Arm A vs Drug Arm B; Difference in change in VAS-A; Test type: Other; p = 0.5351, t-test, 2 sided — The a priori threshold for statistical significance was < 0.05

9. Secondary Outcome: Eyelid Edema Score
Description: Physician-assessed grading of eyelid edema. Score range: 0 to 4; higher numbers indicating more severe swelling.
Time Frame: Post-operative day 7
Population: Participants who completed the intervention.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Drug Arm A | Drug Arm B
Number analyzed (Participants) | 65 | 65
score on a scale | 0 [0 to 2] | 0 [0 to 2]
Statistical Analysis 1: Comparison: Drug Arm A vs Drug Arm B; Test type: Other; p = 0.378, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance was < 0.05

10. Secondary Outcome: Ecchymosis Score
Description: Physician-assessed grading of periorbital ecchymosis extension. Score range: 0 to 4; higher numbers indicating more severe ecchymosis.
Time Frame: Post-operative day 7
Population: Participants who completed the intervention.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Drug Arm A | Drug Arm B
Number analyzed (Participants) | 65 | 65
score on a scale | 0 [0 to 4] | 0 [0 to 4]
Statistical Analysis 1: Comparison: Drug Arm A vs Drug Arm B; Test type: Other; p = 0.195, Wilcoxon (Mann-Whitney) — The a priori threshold for statistical significance was < 0.05

11. Secondary Outcome: Subconjunctival Hemorrhage Score
Description: Physician-assessed grading of subconjunctival hemorrhage. Score range: 0 to 2; higher numbers indicating more severe hemorrhage.
Time Frame: Post-operative day 7
Population: Participants who completed the intervention.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Drug Arm A | Drug Arm B
Number analyzed (Participants) | 65 | 65
score on a scale | 0 [0 to 1] | 0 [0 to 2]
Statistical Analysis 1: Comparison: Drug Arm A vs Drug Arm B; Test type: Other; p = 0.682, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Up 4 weeks pre-procedure through post-operative follow-up (up to an average of 12 months following procedure)
Arm/Group | Drug Arm A | Drug Arm B
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/65
Other Adverse Events (participants affected / at risk) | 0/65 | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT03584152/Prot_000.pdf
  • Statistical Analysis Plan (2025-11-11): https://cdn.clinicaltrials.gov/large-docs/52/NCT03584152/SAP_001.pdf